CLINICAL TRIAL: NCT01260974
Title: Pilot Study: Efficacy of Caspofungin for Antifungal Prophylaxis for Selected High Risk Liver Transplant Patients
Brief Title: Caspofungin as Prophylaxis in High Risk Liver Transplantation Recipients
Acronym: CPHRLTX
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera di Padova (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Prof. Umberto Cillo, Director of the Hepatobiliary Surgery and Liver Transplantation Unit, Azienda Ospedaliera di Padova
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1768P; 2008-007950-36 (EudraCT Number)
Record Dates: First submitted 2010-12-15; First posted 2010-12-16 (Estimated); Last update posted 2012-07-18 (Estimated); Status verified 2012-07

CONDITIONS: Fungemia; Mycoses
Keywords: Invasive fungal infections; Liver Transplantation; Organ Transplantation; Mycoses; Fungus Diseases; Antifungal Agents; Invasive Mycosis
MeSH Terms: conditions — Fungemia; Mycoses; Invasive Fungal Infections | interventions — Caspofungin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Caspofungin (Experimental): Study group
  Interventions: Drug: Caspofungin

INTERVENTIONS:
Drug: Caspofungin — 50mg/dd for 21dd, starting within 24h from Liver Transplantation.
  Other Names: Cancidas

SUMMARY:
The aim of the study is to determine viable use of caspofungin in post-OLTx patients, and to demonstrate in particular the effectiveness, understood as the ability to reduce the incidence of invasive fungal infections, and to assess the ability to reduce the risk and incidence of side effects (toxicity) which may arise in transplant patients treated with other drugs, especially in individuals recognized as high risk (e.g. renal failure).

DETAILED DESCRIPTION:
The prophylactic use of anti-fungal drugs is crucial in order to decrease the incidence of invasive fungal infections in transplantation patients.

Invasive fungal infections (IFI) ---organ-related or systemic infections--- are in fact one of the most important causes of morbidity and mortality in patients undergoing solid organ transplantation (respectively, 70% and 100%).

The rationale of the proposed study is to evaluate a new protocol for the prevention of IFIs through the use of a newly introduced anti-fungal, caspofungin (commercial name: Cancidas), to be used for primary prophylaxis of fungal infections post-OLTx and to compare to drugs already in use (eg. amphotericin B, fluconazole), until 21 days after liver transplantation.

The aim of this study is determine viable use of caspofungin in post-OLTx patients, and to demonstrate in particular the effectiveness, understood as the ability to reduce the incidence of invasive fungal infections, and to assess the ability to reduce the risk and incidence of side effects (toxicity) which may arise in transplant patients treated with other drugs, especially in individuals recognized as high risk (e.g. renal failure).

The possibility of reducing the risk of fungal infections in liver transplant patients (usually between 7 and 42%) is therefore an important clinical goal.

ELIGIBILITY:
Inclusion Criteria:

* patients shortlisted for liver transplantation
* negative pregnancy test for fertile female patients 7 days prior enrollment
* patients who can adequately communicate with study responsibles, who can understand and answer to protocol requirements

At least one of the following criteria:

* MELD score ≥25
* liver transplantation for acute liver failure
* liver re-transplantation
* fever without bacterial or viral infection
* biliodigestive
* re-laparatomy after LTx
* post LTx pancreatitis
* post LTx dialysis or renal insufficiency

Exclusion Criteria:

* Patients enrolled in other clinical trial or those having received other experimental drugs 4 weeks prior to enrollment
* Patients with a known fungal infection (based on the EORTC/MSG criteria)
* Patients with history of hypersensitivity to the drug, or other counterindications
* Patients with a diagnosed Severe Hepatic insufficiency (CTP >9)
* Physical or hematochemical alterations
* Clinically relevant psychological alterations in the 2 weeks preceding enrollment such as to interfere, in the researchers opinion, with the goal of the study
* Patients being treated with Ciclosporin A

Subjects being removed from the trial shall be replaced.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2009-05; Primary Completion 2012-11 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Invasive Fungal Infection Free follow-up | 1 month
  Invasive Fungal Infection free control 1 month after beginning treatment.

SECONDARY OUTCOMES:
Tolerance to treatment. | 3 months
  Tolerance to treatment, with major focus on nephrotoxicity.
Study group mortality | 3 months
  Assessment of study group mortality, compared to control
Study group morbidity | 3 months
  Assessment of study group morbidity, compared to control
Invasive Fungal Infection-free percentage of study group | 1 month
  Invasive Fungal Infection-free percentage of study group, evaluated at 1 month from beginning of study and assessment of mortality and morbidity in the control group

CONTACTS AND LOCATIONS:
Overall Officials: Umberto Cillo, MD, Principal Investigator — Azienda Ospedaliera Universitaria di Padova; Daniele Neri, MD, Principal Investigator — Azienda Ospedaliera Universitaria di Padova
Locations (1):
- Azienda Ospedaliera di Padova, Padua, Padova, Italy

REFERENCES:
- See also: Hepatobiliary surgery and Liver Transplantation Unit, University Hospital of Padua (Italy) — http://www.fegatochirurgia.com/